CLINICAL TRIAL: NCT00025246
Title: A Phase II Study of Adjuvant STI571 (Gleevec TM) Therapy in Patients Following Completely Resected High-risk Primary GastroIntestinal Stromal Tumor (GIST)
Brief Title: Imatinib Mesylate in Treating Patients With Gastrointestinal Stromal Tumor That Has Been Completely Removed During Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03079; ACOSOG-Z9000; U10CA076001 (NIH); CDR0000068942 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-01

CONDITIONS: Gastrointestinal Stromal Tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

ARMS (1):
- Treatment (imatinib mesylate) (Experimental): Patients receive oral imatinib mesylate daily beginning within 84 days of surgical resection. Treatment continues for 1 year in the absence of disease recurrence or unacceptable toxicity.
  Interventions: Drug: imatinib mesylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: imatinib mesylate — Given orally
  Other Names: CGP 57148; Gleevec; Glivec
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well imatinib mesylate works in treating patients with gastrointestinal stromal tumor that was completely removed during surgery. Imatinib mesylate may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To ascertain whether patients with completely resected high-risk primary GIST who undergo adjuvant treatment with STI571 have prolonged survival compared to historical controls.

SECONDARY OBJECTIVES:

I. To determine the 2 and 5-year prevalence of recurrence in patients treated with adjuvant STI571 following complete resection of high-risk primary GIST.

II. To obtain from patients with GIST: tumor tissue (before therapy with STI571 and at the time of recurrence), blood specimens (before therapy with STI571), and serum specimens (before therapy with STI571, after completing therapy with STI571, and at the time of recurrence) for scientific correlative analyses.

III. To assess the toxicity of oral STI571 therapy when used in the adjuvant setting.

OUTLINE:

Patients receive oral imatinib mesylate daily beginning within 84 days of surgical resection. Treatment continues for 1 year in the absence of disease recurrence or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have an ECOG/Zubrod performance status of ≤ 2
* Patient must have a diagnosis of high-risk primary GIST; NOTE: High risk is defined as tumor size ≥ 10 cm in maximum dimension, or the presence of tumor rupture before or during surgery, intraperitoneal hemorrhage or multifocal (< 5) intraperitoneal tumors
* Patient must have undergone complete gross resection (includes R0 [negative microscopic margins] and R1 [positive microscopic margins] resections) of a primary GIST within 70 days prior to registration
* Patient must have a histologic diagnosis of GIST that is confirmed by central pathology review
* Patient's tumor must stain positive for the Kit receptor tyrosine kinase on immunohistochemistry as determined by the central pathologist using the Dako (Dako Corp., Carpinteria, CA) anti-CD 117 antibody
* Patient must have a chest x-ray completed within 28 days prior to registration
* Patient must have a post-operative CT scan with IV and PO contrast or MRI with contrast (if allergic to CT contrast) of abdomen and pelvis within 28 days prior to registration
* Creatinine ≤ 1.5 times the institution ULN
* WBC ≥ 2,000/mm^3
* Platelet ≥ 100,000/mm^3
* Total bilirubin ≤ 1.5 times the institution ULN
* AST and ALT ≤ 2.5 times the institution ULN
* Female of childbearing potential must have negative serum pregnancy test
* Patient or the patient's legally acceptable representative must provide a signed and dated written informed consent prior to registration and any study related procedures
* If patient is a cancer survivor, each of the following criteria must apply:

  * Patient has undergone potentially curative therapy for all prior malignancies,
  * No evidence of any prior malignancies for at least 5 years with no evidence of recurrence (except for effectively treated basal cell or squamous carcinoma of the skin, carcinoma in-situ of the cervix that has been effectively treated by surgery alone, or lobular carcinoma in-situ of the ipsilateral or contralateral breast treated by surgery alone)
  * Patient is deemed by their treating physician to be at low risk for recurrence from prior malignancies

Exclusion Criteria:

* Patient has received post-operative chemotherapy
* Patient has received post-operative radiation therapy
* Patient has received post-operative investigational treatment
* Patient has received prior therapy with STI571
* Patient has had an active infection requiring antibiotics within 14 days prior to registration
* Patient has objective evidence of residual disease on the post-operative CT scan or MRI of the abdomen or pelvis
* Patient, if female and breastfeeding; NOTE: It is not known whether STI571 or its metabolites are excreted in human milk; however, in lactating female rats administered 100 mg/kg, a dose approximately equal to the maximum clinical dose of 800 mg/day based on body surface area, STI571 and/or its metabolites were extensively excreted in milk; it is estimated that approximately 1.5% of a maternal dose is excreted into milk, which is equivalent to a dose to the infant of 30% the maternal dose per unit body weight; because many drugs are excreted in human milk and because of the potential for serious adverse reactions in nursing infants, women should be advised against breastfeeding while taking STI571
* Patient has New York Heart Association class 3 or 4 cardiac disease
* Patient is taking full dose warfarin; NOTE: The use of mini-dose warfarin (1 mg orally per day) for prevention of central line-associated deep venous thrombosis is permitted

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2001-09; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Determination whether patients with completely resected high-risk primary GIST who undergo adjuvant treatment with imatinib mesylate have prolonged survival compared to historical controls | Up to 5 years

SECONDARY OUTCOMES:
Prevalence of recurrence free survival | 2 years
  Marginal point and two-sided 95% (pointwise) confidence bands, based on Kaplan-Meier estimator will be produced.
Prevalence of recurrence | 5 years
  Marginal point and two-sided 95% (pointwise) confidence bands, based on Kaplan-Meier estimator will be produced.
Overall survival | Up to 5 years
  Marginal point and two-sided 95% (pointwise) confidence bands, based on Kaplan-Meier estimator will be produced.
Toxicities, graded according to the National Cancer Institute Common Toxicity Criteria | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Ronald DeMatteo, Principal Investigator — American College of Surgeons
Locations (1):
- American College of Surgeons Oncology Group, Durham, North Carolina, United States

REFERENCES:
- [Derived] DeMatteo RP, Ballman KV, Antonescu CR, Corless C, Kolesnikova V, von Mehren M, McCarter MD, Norton J, Maki RG, Pisters PW, Demetri GD, Brennan MF, Owzar K; American College of Surgeons Oncology Group (ACOSOG) Intergroup Adjuvant GIST Study Team for the Alliance for Clinical Trials in Oncology. Long-term results of adjuvant imatinib mesylate in localized, high-risk, primary gastrointestinal stromal tumor: ACOSOG Z9000 (Alliance) intergroup phase 2 trial. Ann Surg. 2013 Sep;258(3):422-9. doi: 10.1097/SLA.0b013e3182a15eb7. PMID 23860199